CLINICAL TRIAL: NCT02564471
Title: Effect of Antimalarial Drugs on the Immune Response to Rabies Vaccine for Post-exposure Prophylaxis. A Randomized, Open Label, Trial in Healthy US Adults Age 18-60 Years
Brief Title: Effect of Antimalarial Drugs to Rabies Vaccine for Post-exposure Prophylaxis.
Acronym: MALRAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Kansas State University (Other)
Responsible Party: Principal Investigator, Timothy Endy, MD MPH, Chair, Department of Microbiology and Immunology, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 790117
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies | interventions — Chloroquine; chloroquine diphosphate; atovaquone, proguanil drug combination; Doxycycline; Rabies Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Chloroquine (Experimental): Chloroquine Phosphate tablet for oral administration 500 mg chloroquine phosphate (equivalent to 300 mg base)
  Interventions: Drug: Chloroquine; Biological: Rabies Vaccine
- Atovaquone and Proguanil (Malarone) (Experimental): Malarone tablet for oral administration 250 mg atovaquone and 100 mg proguanil hydrochloride.
  RabAvert rabies vaccine, at least 2.5 IU of rabies antigen.
  Interventions: Drug: Atovaquone and Proguanil; Biological: Rabies Vaccine
- Doxycycline (Experimental): Doxycycline hyclate tablet for oral administration, contains specially coated pellets of doxycycline hyclate equivalent to 100 mg of doxycycline.
  RabAvert rabies vaccine, at least 2.5 IU of rabies antigen.
  Interventions: Drug: Doxycycline; Biological: Rabies Vaccine
- Rabies (Active Comparator): RabAvert rabies vaccine, at least 2.5 IU of rabies antigen.
  Interventions: Biological: Rabies Vaccine

INTERVENTIONS:
Drug: Chloroquine — FDA approve dosing schedule
  Other Names: Chloroquine Phosphate
  Arms: Chloroquine
Drug: Atovaquone and Proguanil — FDA approve dosing schedule
  Other Names: Malarone
  Arms: Atovaquone and Proguanil (Malarone)
Drug: Doxycycline — FDA approve dosing schedule
  Other Names: Doxycycline Hyclate
  Arms: Doxycycline
Biological: Rabies Vaccine — FDA approve dosing schedule
  Other Names: RabAvert

SUMMARY:
This is an exploratory trial to evaluate the effect of antimalarial drugs on the immune response generated by rabies vaccine when administered for post-exposure prophylaxis. This study will use the FDA approved post-exposure prophylaxis vaccine regimen (without rabies immune globulin) in the presence or absence of an FDA-approved malaria chemoprophylaxis regimen.

DETAILED DESCRIPTION:
Rabies is present on all continents where U.S. military personnel deploy, including countries where malaria is also endemic and where U.S. military personnel are required to take malaria prophylaxis. Rabies post-exposure prophylaxis in unvaccinated individuals who are not on malaria prophylaxis consists of four, 1.0-mL intramuscular (IM) injections of the purified chick embryo cell (PCECV) rabies vaccine on days 0, 3, 7, and 14. The current Advisory Committee on Immunization Practices (ACIP) guidelines recommend that exposed persons who are taking malaria prophylaxis should receive a fifth dose of rabies vaccine 28 days after the exposure. These guidelines do not differentiate between drugs used for malaria prophylaxis This study will administer the post-exposure regimen to volunteers from a US population of military age who are taking one of three malaria prophylaxis regimens or no malaria prophylaxis. The goal of this study is to asses if individuals on malaria prophylaxis achieve the required rabies titer after completion of the four dose regimen.

Obtaining rabies vaccine and rabies immune globulin in a deployed setting can be challenging. A full understanding of the requirements for protecting exposed individuals is necessary for appropriate decision making in a resource-constrained environment.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent form.
2. Willing to comply with all study procedures and be available for the duration of the study.
3. Male or female, aged ≥ 18 to ≤ 60 years on day of inclusion.
4. In good general health based on medical history and physical exam

Exclusion Criteria:

1. Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination.
2. Participation in the 4 weeks preceding the first trial vaccination, or planned participation during the present trial period, in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
3. Previous history of receiving the rabies vaccine.
4. Previous history of receiving rabies immune globulin.
5. Any major psychiatric disorder, such as severe depression, severe anxiety disorder, psychosis, schizophrenia, other major psychiatric disorders, or seizures. History of mild depression or anxiety disorder that are well controlled are not exclusion criteria.
6. Use of any immunosuppressive drug at the time of the study or 30 days previously. Topical steroids will not be considered an immunosuppressive drug and their use will not be considered an exclusion criteria.
7. Any immunosuppressive disorder, such as HIV infection, common variable immunodeficiency, active cancers or chemotherapy.
8. History of renal insufficiency or requiring dialysis.
9. Have any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
10. Identified as an employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employee or the Investigator.
11. Previous adverse reaction to any of the antimalarial drugs used in this study.

Temporary Exclusion Criteria: Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on day 0.. A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided. If the delay for the febrile illness exceeds the window between screening and vaccination, or if deemed necessary by the investigator, a prospective subject may be re-screened once the fever has resolved.

Recent or scheduled receipt of any vaccine 4 weeks prior to day 0.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Endy, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- State University of New York, Upstate Medical University (SUNY-UMU), Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Endy TP, Keiser PB, Cibula D, Abbott M, Ware L, Thomas SJ, Polhemus ME. Effect of Antimalarial Drugs on the Immune Response to Intramuscular Rabies Vaccination Using a Postexposure Prophylaxis Regimen. J Infect Dis. 2020 Mar 2;221(6):927-933. doi: 10.1093/infdis/jiz558. PMID 31743394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults aged 18 to 60 were recruited from 11-Nov-2016 to 07-Jun-2018 in and around the study site in Syracuse, New York
Groups:
- Atovaquone and Proguanil (Malarone): Malarone tablet for oral administration 250 mg atovaquone and 100 mg proguanil hydrochloride.
  RabAvert rabies vaccine, at least 2.5 IU of rabies antigen.
  Atovaquone and Proguanil: FDA approve dosing schedule
  Rabies Vaccine: FDA approve dosing schedule
- Doxycycline: Doxycycline hyclate tablet for oral administration, contains specially coated pellets of doxycycline hyclate equivalent to 100 mg of doxycycline.
  RabAvert rabies vaccine, at least 2.5 IU of rabies antigen.
  Doxycycline: FDA approve dosing schedule
  Rabies Vaccine: FDA approve dosing schedule
Period: Overall Study
Arm/Group | Chloroquine | Atovaquone and Proguanil (Malarone) | Doxycycline | Rabies
Started | 25 | 26 | 27 | 25
Completed | 22 | 23 | 24 | 25
Not Completed | 3 | 3 | 3 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Group 1: 1 subject excluded from analysis due to presence of rabies antibody titer at baseline; 1 excluded due to use of steroids during the study.
  Group 3: 1 subject excluded from analysis due to presence of rabies antibody titer at baseline
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroquine | Atovaquone and Proguanil (Malarone) | Doxycycline | Rabies | Total
Number analyzed (Participants) | 20 | 23 | 23 | 25 | 91
Age, Categorical [Count of Participants; unit: Participants] — Population: Group 1: 3 subjects withdrew; 1 subject was excluded from analysis due to presence of rabies antibody titer at baseline; 1 subject was excluded due to use of steroids during the study.
  Group 2: 3 subjects withdrew. Group 3: 3 subjects withdrew; 1 subject was excluded from analysis due to presence of rabies antibody titer at baseline
  Participants
    <=18 years | 1 | 0 | 1 | 0 | 2
    Between 18 and 65 years | 19 | 23 | 22 | 25 | 89
    >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 13 | 11 | 52
  Male | 8 | 7 | 10 | 14 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 0 | 6
  Not Hispanic or Latino | 19 | 20 | 21 | 25 | 85
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 5 | 10
  White | 18 | 20 | 22 | 18 | 78
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 23 | 23 | 25 | 91
Participants with data available at both baseline and post baseline assessments [Number; unit: participants] | 20 | 23 | 23 | 25 | 91

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) 14 Days Post Fourth Dose Post Exposure Prophylaxis (PEP) With Purified Chick Embryo Cell Vaccine (PCECV) in Each Malaria Prophylaxis Group Compared to Control to Determine if a Fifth Dose of PEP Would Add Value
Description: Chloroquine, Atovaquone and Proguanil (Malarone) and Doxycycline Groups received antimalarial up to day 14 and rabies vaccinations on day 14, 17, 21, and 28 (dose 4). Rabies Group received the rabies vaccination on days 0, 3,7 and 14 (dose 4). Rabies virus-specific serum antibody neutralization assay was used to measure rabies virus antibodies, using the rapid fluorescent foci inhibition test (RFFIT). A titer of >0.5 IU/ml against rabies virus as protective. Descriptive analyses were based on samples taken 14 days after dose 4, (e.g., at 6 weeks for Chloroquine, Atovaquone and Proguanil (Malarone) and Doxycycline Arms and at 4 weeks for Rabies Arm).
Time Frame: 6 weeks for Chloroquine, Atovaquone and Proguanil (Malarone) and Doxycycline Groups and at 4 weeks for Rabies Group
Population: Group 1: 1 subject was excluded from analysis due to presence of rabies antibody titer at baseline, 1 was excluded due to use of steroids during the study; Group 2: 1 subject completed primary endpoint but did not complete the study; Group 3: 1 subject was excluded from analysis due to presence of rabies antibody titer at baseline
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/ml
Arm/Group | Chloroquine | Atovaquone and Proguanil (Malarone) | Doxycycline | Rabies
Number analyzed (Participants) | 20 | 24 | 23 | 25
IU/ml | 3.45 (1.62) | 7.95 (0.81) | 8.51 (0.94) | 10.26 (0.66)

2. Secondary Outcome: GMT Over Protective Titer Prior to Third Dose of PCECV
Description: Chloroquine, Atovaquone and Proguanil (Malarone) and Doxycycline Groups received antimalarial up to day 14 and rabies vaccinations on day 14, 17, 21 (dose 3), and 28 (dose 4). Rabies Group received the rabies vaccination on days 0, 3, 7 (dose 3) and 14 (dose 4). For Chloroquine, Malarone and Doxycycline Groups, samples were taken on days 0, 21, 28 and 56. For Rabies Group, samples were taken on days 0, 7, 14 and 42. Rabies virus-specific serum antibody neutralization assay was used to measure rabies virus antibodies, using the rapid fluorescent foci inhibition test (RFFIT). A titer of >0.5 IU/ml against rabies virus as protective.
Time Frame: 21 days for Chloroquine, Atovaquone and Proguanil (Malarone) and Doxycycline Groups and 7 days for Rabies Arm
Population: Group 1: 1 subject completed all doses of vaccine but did not complete the study; Group 2: 2 subjects completed all doses of vaccine but did not complete the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/ml
Arm/Group | Chloroquine | Atovaquone and Proguanil (Malarone) | Doxycycline | Rabies
Number analyzed (Participants) | 21 | 25 | 23 | 25
IU/ml | 0.14 (0.62) | 0.11 (0.40) | 0.16 (0.72) | 0.17 (1.15)

3. Secondary Outcome: GMT Over Protective Titer Prior Fourth Dose of PCECV
Description: as for outcome 2
Time Frame: 28 days for Chloroquine, Atovaquone and Proguanil (Malarone) and Doxycycline Groups and 14 days for Rabies Arm
Population: Group 1: 1 subject received all doses but did not complete the study; Group 2: 2 subjects received all doses but did not complete the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/ml
Arm/Group | Chloroquine | Atovaquone and Proguanil (Malarone) | Doxycycline | Rabies
Number analyzed (Participants) | 21 | 25 | 23 | 25
IU/ml | 4.15 (289) | 6.45 (1.39) | 7.04 (2.71) | 6.98 (1.12)

4. Secondary Outcome: GMT Over Protective Titer 28 Days Post Fourth Dose of PCECV
Description: Chloroquine, Atovaquone and Proguanil (Malarone) and Doxycycline Groups received antimalarial up to day 14 and rabies vaccinations on day 14, 17, 21 (dose 3), and 28 (dose 4). Rabies Group received the rabies vaccination on days 0, 3,7 (dose 3) and 14 (dose 4). For Chloroquine, Malarone and Doxycycline Groups, samples were taken on days 0, 21, 28 and 56. For Rabies Group, samples were taken on days 0, 7, 14 and 42. Rabies virus-specific serum antibody neutralization assay was used to measure rabies virus antibodies, using the rapid fluorescent foci inhibition test (RFFIT). A titer of >0.5 IU/ml against rabies virus as protective.
Time Frame: Up to 8 weeks for Chloroquine, Atovaquone and Proguanil (Malarone) and Doxycycline Groups and up to 6 weeks for Rabies Arm
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/ml
Arm/Group | Chloroquine | Atovaquone and Proguanil (Malarone) | Doxycycline | Rabies
Number analyzed (Participants) | 20 | 23 | 23 | 25
IU/ml | 2.3 (1.53) | 4.96 (0.78) | 5.18 (1.14) | 6.87 (1.04)

ADVERSE EVENTS:
Time Frame: 8 weeks from Chloroquine, Malarone/Atovaquone, Doxycyline groups, 6 weeks for rabies control group.
Groups:
- Doxyclycline: Doxycycline hyclate tablet for oral administration, contains specially coated pellets of doxycycline hyclate equivalent to 100 mg of doxycycline.
  RabAvert rabies vaccine, at least 2.5 IU of rabies antigen.
  Doxycycline: FDA approve dosing schedule
  Rabies Vaccine: FDA approve dosing schedule
Arm/Group | Chloroquine | Atovaquone and Proguanil (Malarone) | Doxyclycline | Rabies
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 17/25 | 22/26 | 19/27 | 19/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Chloroquine (N=25) | Atovaquone and Proguanil (Malarone) (N=26) | Doxyclycline (N=27) | Rabies (N=25)
Abdominal Pain (Gastrointestinal disorders) | 4 | 3/23 | 0/23 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4/20 | 4 | 6/23 | 4
Injection site reaction (General disorders) | 9 | 11 | 10 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 3 | 1
Flu like symptoms (General disorders) | 3 | 1 | 2 | 2
Upper Respiratory Infection (Infections and infestations) | 1 | 4 | 2 | 4
Headache (Nervous system disorders) | 4 | 9 | 7 | 3
Fatigue (General disorders) | 1 | 1 | 4 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 5 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 0
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 — Sunburn

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT02564471/Prot_001.pdf
  • Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT02564471/SAP_000.pdf
  • Informed Consent Form (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT02564471/ICF_002.pdf